CLINICAL TRIAL: NCT00104962
Title: Phase I Study of CC-5013 (Lenalidomide NSC# 703813) in Pediatric Patients With Relapsed/Refractory Solid Tumors or Myelodysplastic Syndrome
Brief Title: Lenalidomide in Treating Young Patients With Relapsed or Refractory Solid Tumors or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01820; NCI-2012-01820 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL0319; NCI-P6553; CDR0000413700; NCI-06-C-0052; ADVL0319 (Other: COG Phase I Consortium); ADVL0319 (Other: CTEP); U01CA097452 (NIH); NCT00269711 (obsolete NCT alias)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2012-12

CONDITIONS: Childhood Myelodysplastic Syndromes; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Ringed Sideroblasts; Refractory Cytopenia With Multilineage Dysplasia; Secondary Myelodysplastic Syndromes; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Lenalidomide

ARMS (1):
- Treatment (lenalidomide) (Experimental): Patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid

SUMMARY:
This phase I trial is studying the side effects and best dose of lenalidomide in treating young patients with relapsed or refractory solid tumors or myelodysplastic syndromes. Lenalidomide may stop the growth of solid tumors or myelodysplastic syndromes by blocking blood flow to the cancer. It may also stimulate the immune system in different ways and stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of lenalidomide in pediatric patients with relapsed or refractory solid tumors.

II. Determine the toxic effects of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine, preliminarily, the feasibility of administering this drug to pediatric patients with relapsed or refractory myelodysplastic syndromes.

II. Determine, preliminarily, the antitumor activity of this drug in both patient populations.

III. Determine immunologic changes in patients treated with this drug.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to diagnosis (solid tumor vs myelodysplastic syndromes [MDS]).

Patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients with solid tumors receive escalating doses of lenalidomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Patients with MDS receive a fixed dose (do not undergo dose escalation) of lenalidomide. After completion of study treatment, patients are followed annually.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Histologically confirmed solid tumor

    * No brain tumors
  * Myelodysplastic syndromes (MDS)

    * No refractory anemia with excess blasts in transformation or other forms of acute myeloid leukemia (AML)
    * No FAB diagnosis of refractory anemia with excess blasts in transition and other forms of AML
    * Newly diagnosed MDS with chromosome 5q abnormalities
* Relapsed or refractory disease including relapse after stem cell transplantation
* Measurable or evaluable disease (solid tumor patients only)
* No known curative or life-prolonging therapy exists
* No bone marrow involvement by tumor (solid tumor patients only)
* No CNS tumors
* Performance status - Karnofsky 50-100% (for patients > 10 years of age)
* Performance status - Lansky 50-100% (for patients ≤ 10 years of age)
* Absolute neutrophil count ≥ 1,000/mm^3 (for patients with solid tumors)
* Platelet count ≥ 100,000/mm^3 (30,000 for patients with MDS)

  * Only patients with MDS may receive transfusions to support platelet counts
* Hemoglobin ≥ 8.0 g/dL (transfusions allowed)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 110*
* Albumin ≥ 2 g/dL
* Creatinine clearance OR radioisotope glomerular filtration rate ≥ 70 mL/min
* Creatinine based on age as follows:

  * Creatinine ≤ 0.8 mg/dL (for patients ≤ 5 years of age)
  * Creatinine ≤ 1 mg/dL (for patients 6 to 10 years of age)
  * Creatinine ≤ 1.2 mg/dL (for patients 11 to 15 years of age)
  * Creatinine ≤ 1.5 mg/dL (for patients over 15 years of age)
* No parent or sibling with a known history of venous thrombosis before the age of 50 OR arterial thrombosis before the age of 40
* No thromboembolic event except catheter-related thrombosis
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception 4 weeks before, during, and for ≥ 4 weeks after completion of study treatment
* Body surface area ≥ 0.4m^2
* No uncontrolled infection
* No active graft-vs-host disease from prior stem cell transplant or rescue
* Recovered from prior immunotherapy
* At least 1 week since prior biologic agents
* At least 1 week since prior hematologic growth factors (2 weeks for pegfilgrastim)
* At least 3 months since prior stem cell transplant or rescue (without total body irradiation [TBI])
* Prior thalidomide allowed
* No other concurrent immunotherapy
* No other concurrent biologic therapy
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent chemotherapy
* Concurrent dexamethasone allowed provided the dose has been either decreasing or stable for the past 7 days
* See Biologic therapy
* Recovered from prior radiotherapy
* At least 2 weeks since prior local palliative (small port) radiotherapy
* At least 6 months since prior TBI, craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* No concurrent radiotherapy
* No other concurrent investigational drugs or agents
* No other concurrent anticancer agents

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2005-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of lenolidomide defined as the maximum dose at which fewer than one-third of patients experience DLT | 28 days
  Graded using the CTCAE version 3.0.

SECONDARY OUTCOMES:
Overall response assessed using RECIST criteria | Up to 30 days after completion of study treatment
  A patient will be considered to have responded if she or he demonstrates either a bone marrow or cytogenetic response. Each patient will be classified according to the maximum response of the two criteria, where the classification from maximum to minimum will be: CR, PR or nonresponse.
Adverse events defined using the NCI CTCAE version 3.0 | Up to 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Berg, Principal Investigator — COG Phase I Consortium
Locations (1):
- COG Phase I Consortium, Arcadia, California, United States

REFERENCES:
- [Derived] Berg SL, Cairo MS, Russell H, Ayello J, Ingle AM, Lau H, Chen N, Adamson PC, Blaney SM. Safety, pharmacokinetics, and immunomodulatory effects of lenalidomide in children and adolescents with relapsed/refractory solid tumors or myelodysplastic syndrome: a Children's Oncology Group Phase I Consortium report. J Clin Oncol. 2011 Jan 20;29(3):316-23. doi: 10.1200/JCO.2010.30.8387. Epub 2010 Dec 13. PMID 21149673